CLINICAL TRIAL: NCT04840706
Title: Open-Label Prospective Study Comparing Long-Term Outcome With or Without High-flow Nasal Cannula AirvoTM in Patients With Stable Hypercapnic COPD
Brief Title: Open-Label Prospective Study Comparing Long-Term Outcome With or Without HFNC in Patients With Stable Hypercapnic COPD
Acronym: MyAirvo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was not possible to achieve recruitment target
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Tarja Saaresranta, Principal Investigator, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MyAirvo
Record Dates: First submitted 2021-04-09; First posted 2021-04-12 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Airvo (Active Comparator): Patients allocated to use Airvo device
  Interventions: Device: HFNC Airvo
- Control (Placebo Comparator): Patients not using Airvo, standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Device: HFNC Airvo — HFNC device (Airvo) long-term use in in stabile hypercapnic COPD patients, who are non-compliant to NIV after an acute exacerbation of COPD
  Arms: Airvo
Other: Standard care — No HFNC treatment
  Arms: Control

SUMMARY:
The aims of the study are to compare long-term one-year outcome with or without AirvoTM in stabile hypercapnic COPD patients, who are non-compliant to NIV after an acute exacerbation of COPD.

DETAILED DESCRIPTION:
When compared to NIV, much less experience is available from clinical studies on HFNC therapy. Until now, few studies have investigated the effect of HFNC therapy on hypercapnic COPD patients and the number of patients recruited in these studies is limited. AirvoTM therapy could be good choice of treatment for those COPD patients that are not compliant to NIV but need treatment for hypercapnia in order to reduce COPD exacerbations and enhance QOL.The aims of the study are to compare long-term one-year outcome with or without AirvoTM in stabile hypercapnic COPD patients, who are non-compliant to NIV after an acute exacerbation of COPD.

ELIGIBILITY:
Inclusion Criteria:COPD patients 1) with at least two acute moderate or severe exacerbations during past 12 months, 2) who at the follow-up visit one month after an acute severe exacerbation of COPD are hypercapnic (capillary pCO2 >6.5 kPa) and not willing to use NIV or have used it less than 4 h/d during the last month despite optimal settings prescribed by an experienced pulmonologist, or if a patient at the follow-up one month after a severe exacerbation is hypercapnic and is willing to try NIV (initiated at the follow-up visit, not at the ward), but then uses it less than 4h/d during the following month. Acute moderate (treated with short acting bronchodilators plus antibiotics and/or oral corticosteroids) and severe (patient requires hospitalization or visits the emergency room) exacerbations of COPD are defined according to the GINA Guidelines (GOLD 2019).

Exclusion Criteria: 1) OSA (diagnosed OSA or high suspicion OSA because of regular snoring, witnessed apneas and daytime sleepiness), 2) neuromuscular or chest wall disease, 3) BMI>35 kg/m2 or 4) a patient is not able to give his/her informed consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
pCO2 | 1 year
  Improvement in daytime capillary pCO2 ≥ 0.5 kPa in the AirvoTM group compared to the standard care group
Acute exacerbation rate | 1 year
  decrease in acute exacerbation (moderate or severe) rate of COPD in AirvoTM group compared to the previous 12 months before entering the study and standard care group

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland